CLINICAL TRIAL: NCT01953952
Title: Randomized Phase II Trial of Transoral Endoscopic Head And Neck Surgery Followed by Risk-Based IMRT and Weekly Cisplatin Versus IMRT and Weekly Cisplatin for HPV Negative Oropharynx Cancer
Brief Title: Radiation Therapy and Cisplatin With or Without Surgery in Treating Patients With Stage III-IV Oropharyngeal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1221; NCI-2013-00939 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG 1221 (Other: Radiation Therapy Oncology Group); RTOG-1221 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

ARMS (2):
- Arm I (surgery, risk-based adjuvant therapy) (Experimental): Patients undergo eHNS. Depending on post-operative pathology findings, patients may undergo IMRT QD five days a week for 6 weeks, beginning within 6 weeks after surgery. High-risk patients also receive cisplatin IV on days 1, 8, 15, 22, 29, and 36 during radiation therapy.
  Interventions: Procedure: therapeutic conventional surgery; Radiation: intensity-modulated radiation therapy; Drug: cisplatin; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis
- Arm II (chemoradiotherapy) (Active Comparator): Patients undergo IMRT QD five days a week for 7 weeks. Patients also receive cisplatin IV on days 1, 8, 15, 22, 29, and 36 during radiation therapy.
  Interventions: Radiation: intensity-modulated radiation therapy; Drug: cisplatin; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo transoral eHNS
  Arms: Arm I (surgery, risk-based adjuvant therapy)
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies radiation therapy and cisplatin with or without surgery in treating patients with stage III-IV oropharyngeal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy with radiation therapy may kill more tumor cells. It is not yet known whether radiation therapy and cisplatin are more effective with or without surgery in treating patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if primary treatment with transoral endoscopic head and neck surgery will improve progression free survival (PFS) for patients with human papilloma virus negative (HPV-) oropharyngeal cancer (OPC).

SECONDARY OBJECTIVES:

I. To compare patterns of failure (local-regional relapse versus distant) and survival (overall and progression-free).

II. To determine the safety and efficacy (rate of positive surgical margins) of using transoral robotic surgery for patients with T3 tumors of the tonsil, tongue-base, or glossopharyngeal sulcus.

III. To compare head and neck cancer-specific quality of life (QOL) short-term (< 6 months) and long-term (2 years) relating to swallowing function.

IV. To compare subjective (patient reported) and objective (physiologic) measures of swallowing function short-term and long-term.

V. To assess effect of neck dissection on shoulder function using a validated QOL instrument for patients undergoing neck dissection VI. To assess the correlation of physician derived clinical target volumes (CTV's) with locoregional control or failure.

VII. To determine whether specific molecular profiles are associated with overall or progression-free survival or other clinical endpoints.

VIII. To determine the sensitivity and specificity of pre-treatment computed tomography (CT) scans detecting the presence of lymph node extracapsular extension by examining the surgically dissected lymph nodes.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo transoral endoscopic head and neck surgery (eHNS). Depending on post-operative pathology findings, patients may undergo intensity modulated radiation therapy (IMRT) once daily (QD) five days a week for 6 weeks. High-risk patients also receive cisplatin intravenously (IV) on days 1, 8, 15, 22, 29, and 36 during radiation therapy.

ARM II: Patients undergo IMRT QD five days a week for 7 weeks. Patients also receive cisplatin IV on days 1, 8, 15, 22, 29, and 36 during radiation therapy.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma of the oropharynx, localized to the tonsil, glossopharyngeal sulcus, and tongue-base within 6 weeks (42 days) of registration
* The primary tumor must be resectable through a transoral endoscopic head and neck surgery with anticipation of resection free margins (resection does not require total or subtotal glossectomy or total laryngectomy); specifically, patients must (1) not have trismus, (2) not have interincisor opening less than 2.5 cm, and (3) not have poor transoral exposure of the tumor itself nor surrounding soft-tissue margins, regardless of etiology
* Clinical stage III-IV; T1-2, N1-2b; T3, N0-2b, with only well-lateralized exophytic T3 tumors not approaching within 1 cm of midline, and amenable to transoral eHNS
* p16 protein (p16) negative by immunohistochemistry (documented by the institution's pre-enrollment biomarker screening at a Clinical Laboratory Improvement Amendments [CLIA]-certified lab), defined as absent, weak, and/or only focal nuclear and cytoplasmic staining in less than 70% of the tumor cells
* Appropriate stage for protocol entry, including no distant metastases or adenopathy below the clavicles, based upon the following minimum diagnostic workup:

  * History/physical examination by the treating physician (radiation oncologist, medical oncologist, or head and neck surgeon) within 30 days prior to registration
  * Imaging of the head and neck (CT with contrast, positron emission tomography [PET]/CT, and/or magnetic resonance imaging [MRI]) within 30 days prior to registration; a CT scan with contrast is mandatory (unless contraindicated, e.g. contrast allergy, etc.); note that a PET/CT scan alone (unless performed with contrast) is not sufficient
  * Chest CT scan (with or without contrast) or PET/CT of chest (with or without contrast) within 30 days prior to registration
  * Modified barium swallow (MBS) to assess swallowing function within 30 days prior to registration
  * Preoperative Mallampati assessment as documented by attending surgeon within 30 days prior to registration
* Zubrod performance status 0-1 within 30 days prior to registration
* Absolute neutrophil count (ANC) >= 1,800 cells/mm^3 based upon complete blood count (CBC)/differential
* Platelets >= 100,000 cells/mm^3 based upon CBC/differential
* Hemoglobin >= 8.0 g/dl based upon CBC/differential (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Total bilirubin =< 2 mg/dl
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the upper limit of normal
* Serum creatinine =< 1.5 mg/dl and/or creatinine clearance (CC) >= 50 ml/min; CC can be determined by 24-hour collection or estimated by Cockcroft-Gault formula
* Serum pregnancy test within 14 days prior to registration for women of childbearing potential
* Women of childbearing potential and male participants who are sexually active must practice medically effective contraception during treatment and for 42 days following completion of treatment
* Patient must be able to provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (for example, carcinoma in situ of the breast or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity, defined as follows:

  * > 2 based on the American Society of Anesthesiologists (ASA) physical status classification system
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive; protocol-specific requirements may also exclude immuno-compromised patients
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Prior allergic reaction to cisplatin
* Radiographic evidence of retropharyngeal metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  Estimated for both arms using the Kaplan-Meier method. The distribution will be compared between arms with a one-sided log rank test.

SECONDARY OUTCOMES:
Patterns of local, regional, and distant failure | Up to 5 years
  The cumulative incidence method will be used to estimate local-regional and distant failure rates and the failure rates for the experimental treatment will be compared against the control using a failure specific log rank test.
Overall survival (OS) | Up to 5 years
  Estimated for both arms using the Kaplan-Meier method. The distribution will be compared between arms with a one-sided log rank test.
Rate of grade 4-5 oropharyngeal hemorrhage and involved surgical margin for all patients and patients with selected T3 tumors | Up to 5 years
Objective swallowing function | Up to 2 years
Shoulder function | Up to 2 years
Short-term quality of life: head and neck-specific (swallowing domain and shoulder function) using the M. D. Anderson Dysphagia Inventory (MDADI) | Up to 6 months
  Compared using a two-sample independent t test and paired t test if the comparison is within the experimental arm between different time points. Overall score and change from baseline will be summarized using mean and standard deviation at each time point for each arm. Binary endpoints will be compared using Fisher's exact test.
Long-term quality of life: head and neck-specific (swallowing domain and shoulder function) using the MDADI | At 2 years
  Compared using a two-sample independent t test and paired t test if the comparison is within the experimental arm between different time points. Overall score and change from baseline will be summarized using mean and standard deviation at each time point for each arm. Binary endpoints will be compared using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Floyd C. Holsinger, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States